CLINICAL TRIAL: NCT06250920
Title: Effect of Virtual Reality-Based Visual Training for Myopia Control in Children: a Randomized Controlled Trial
Brief Title: Effect of Virtual Reality-Based Visual Training for Myopia Control in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Jing Yu, Dr, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4.1/20-260/01
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Myopia; Myopia, Progressive
MeSH Terms: conditions — Myopia; Myopia, Degenerative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality-based visual training group (Experimental)
  Interventions: Device: Virtual reality visual training
- Single-Vision Spectacle Group (No Intervention)

INTERVENTIONS:
Device: Virtual reality visual training — Children in intervention group were administered at home under the supervision of parents for 20 minutes per session every day with virtual reality visual training
  Arms: Virtual reality-based visual training group

SUMMARY:
To assess the efficacy and safety of virtual reality-based visual training (VRVT) in myopia control among children.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-13 years old (inclusive), regardless of gender;
2. The spherical equivalent of both eyes after cycloplegia was -3.00D to -0.50D (including);
3. Binocular astigmatism ≤3.00D during screening;
4. Anisometropia (according to spherical equivalent) ≤1.50D during screening;
5. The intraocular pressure of any eye during screening was ≤21mmHg;
6. At the time of screening, the best corrected distance visual acuity of any eye was ≥1.0 or LogMAR≤0;
7. Good binocular stereopsis and stereopsis acuity ≤60 ";
8. The subjects and their legal guardians were willing to participate in the study and signed written informed consent.

Exclusion Criteria:

1. Existing or previous history of ophthalmic organic diseases, ophthalmic surgery, and obvious strabismus after wearing glasses;
2. Using orthokeratology lenses, feeding instrument and other myopia prevention and control methods that may affect the study in the past 6 months;
3. Subjects with poor vestibular function such as motion sickness and seasickness;
4. Any history of diseases or syndromes that may cause severe myopia (e.g., Marfan syndrome, Stickler syndrome, retinopathy of prematurity, etc.); 5, any eye refractive media abnormalities (such as cornea, lens abnormalities, etc.);

6. Long-term use (i.e., more than 7 consecutive days in 1 month or more than 30 days in total in 1 year) of any local or systemic use of anticholinergic/anticholinergic drugs (e.g., atropine, scopolamine, tolacamide, etc.) within 21 days before screening and during the expected period of the study, allowing the use of cycloplegic drops for optometry and other examinations; 7. Severe systemic disease considered by the investigator as not suitable for the study; 8. Participation in other clinical trials within 30 days before screening; 9. Only one eye met the inclusion criteria; 10. Poor compliance, unable to go to medical institutions for treatment on a timely and regular basis as required; 11. Any other circumstances deemed inappropriate by the investigator to participate in the study.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
changes in axial length | baseline and the 3-month follow-up visits

SECONDARY OUTCOMES:
changes in subfoveal choroidal thickness | baseline and the 3-month follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu Z, Zou A, Li L, Wu Y, Cai W, Ma J, Yu J. Effect of virtual reality-based visual training for myopia control in children: a randomized controlled trial. BMC Ophthalmol. 2024 Sep 16;24(1):358. doi: 10.1186/s12886-024-03580-w. PMID 39278928